CLINICAL TRIAL: NCT05039554
Title: Randomized Trial of Acceptance and Commitment Therapy (ACT) and a Care Management App in Primary Care-based Buprenorphine Treatment
Brief Title: Randomized Trial of ACT and a Care Management App in Primary Care-based Buprenorphine Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13325; RM1DA055437 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-09-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Opioid-use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Valera smartphone application (app) alone (Active Comparator): Participants randomized to this cohort will receive the Valera app and will receive a smartphone with network connectivity if necessary.
  Interventions: Other: Valera Smartphone Application
- ACT + Valera app (Experimental): Participants randomized to this cohort will receive both acceptance and commitment therapy (ACT) and the Valera app (and a smartphone with network connectivity if necessary).
  Interventions: Behavioral: Acceptance and commitment therapy; Other: Valera Smartphone Application
- treatment as usual (TAU) (Placebo Comparator): Participants randomized to this cohort will not receive any experimental treatments.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Intervention will be provided over 12 weeks with weekly 1-hour sessions using a group format with the overall goal to foster psychological flexibility. ACT will assist participants to notice their internal triggers; abandon their attempts to manage these triggers via active avoidance (suppression or other control-based strategies including opioid or other substance use) and to make commitments to engage in behaviors consistent with their chosen values or goals (rather than allowing negative thoughts, feelings, or pain symptoms to dictate behavior).
  Other Names: ACT
  Arms: ACT + Valera app
Other: Valera Smartphone Application — For those randomized to a cohort with the Valera app, the app (and cellphones if necessary) will be provided. The app is HIPAA compliant and IRB approved. It consists of 2 components: a participant-facing Smartphone Application and a corresponding online Care Manager Dashboard. Smartphones and internet access will be provided as needed for the 12-week study duration.
  Arms: ACT + Valera app; Valera smartphone application (app) alone
Other: Treatment as Usual — TAU for BUP treatment typically consists of regularly scheduled visits every 1-2 months with primary care physicians and/or nurse care managers in Montefiore primary care settings. During these 15-min follow up visits, providers typically inquire about opioid and other substance use, opioid craving, symptoms of opioid withdrawal, and risk of relapse. In addition, at each visit, urine toxicology tests are conducted and providers review results of prior urine toxicology tests with patients. If opioid or other substance use is ongoing, typically providers will intensify treatment, including increasing the frequency of visits, referring to social workers or mental health providers, recommending self-help groups, and/or recommending outpatient drug treatment programs (e.g., individual and group counseling).
  Other Names: TAU
  Arms: treatment as usual (TAU)

SUMMARY:
The proposed IMPOWR Research Center at Montefiore-Einstein (IMPOWR-ME) will create a multidisciplinary and synergistic program of research to test multimodal treatments that address both chronic pain and opioid use disorder. IMPOWR-ME will generate critical knowledge about the effectiveness, implementation, and cost effectiveness of providing Acceptance and Commitment Therapy and/or a care management smartphone app for individuals in primary care-based buprenorphine treatment. Patients with lived experience with chronic pain and/or opioid use disorder, patient and policy advocates, payors, and health system partners will be engaged in all stages of the research. IMPOWR-ME is well-positioned to become a long-lasting hub for stakeholder-engaged research with multidisciplinary senior and early stage investigators focused on reducing overdose through better treatments for OUD and CP.

DETAILED DESCRIPTION:
Chronic pain (CP) and opioid use disorder (OUD) are leading causes of morbidity and mortality in the United States. Despite being commonly comorbid, there is a striking lack of integrated treatments accessible to people in need. This is particularly true for Black and Hispanic individuals living and seeking care in under-resourced settings like The Bronx, NY, one of the poorest and most racially diverse counties in the U.S. Submitted in response to the HEAL Initiative: Integrative Management of Chronic Pain and OUD for Whole Recovery (IMPOWR) RFA-DA-21-030, the overall goal of this proposal is to create the IMPOWR Research Center at Montefiore/Einstein ("IMPOWR-ME"), in the high-impact county of The Bronx NY. IMPOWR-ME is a synergistic multidisciplinary research center that leverages exceptional research infrastructure in CP and OUD and existing relationships with people living with CP and OUD, advocates, policymakers and payers, and health system stakeholders. The aims of IMPOWR-ME are to: 1) create a robust and sustainable research infrastructure to rigorously test and disseminate integrated and cost-effective evidence-based practices for people with CP and OUD; 2) partner with people with lived experience with CP, OUD, or both, and diverse stakeholders in all stages of the research; and 3) provide opportunities for multidisciplinary early stage investigators to become independent researchers focusing on CP and OUD. This innovative hybrid type 1 effectiveness-implementation trial is proposed to rigorously examine multi-modal evidence-based practices in diverse health care settings and populations of people with comorbid CP and OUD. Specifically, the investigators propose a 2x2 factorial trial to test Acceptance and Commitment Therapy and a care management smartphone app for individuals in primary-care based buprenorphine treatment. Participants will have both CP and OUD or opioid misuse, and specific aims will examine CP, OUD, implementation, and cost-effectiveness outcomes; additional patient-centered outcomes will be driven by people with lived experience. This project improves access to care for Black and Hispanic individuals in under-resourced settings by bringing integrated treatment of CP and OUD to them, and the interventions have high potential for dissemination and sustainability. An innovative program for pilot studies achieves a dual aim of catalyzing stakeholder-driven research and training early stage and new investigators. An exceptional team of investigators and clinical experts focused on CP and OUD, a longstanding history of collaboration with stakeholders and people with lived experience, and a high-impact population make Montefiore-Einstein an ideal site for an IMPOWR research center.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older;
2. English or Spanish proficiency;
3. receiving BUP treatment for OUD for at least 14 days (thus a stabilized BUP dose); and
4. CP with at least moderate pain severity (score greater than or equal to 4 on Pain, Enjoyment of Life and General Activity scale (PEG). Comorbid psychiatric conditions and use of psychotropic medications will be allowed.

Exclusion Criteria:

1. Acute exacerbation of psychiatric conditions precluding the ability to participate in the study (e.g., acute mania, active suicidality/homicidality, psychosis);
2. psychotropic medication changes within the past three months prior to enrollment;
3. CP related to malignancy;
4. received ACT or similar therapeutic intervention in the past;
5. initiated psychotherapy within the past three months;
6. neurocognitive conditions that may prevent participants from accessing telehealth services;
7. current use of a smartphone health platform similar to the Valera app;
8. are unable or unwilling to provide signed consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pain interference | Baseline, 30 days, 12 weeks, 36 weeks
  The primary outcome for pain will be pain-related functional interference, assessed with the Brief Pain Inventory (BPI), pain interference subscale, a nine-item measure that assesses pain related interference with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The total score has demonstrated reliability (e.g., Cronbach's Alpha = 0.86) and validity with chronic pain patients.
Opioid Use | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Opioid use will be measures by the Addiction Severity Index (ASI), which provides an assessment of drug use in the past 30 days, as done in our other studies.

SECONDARY OUTCOMES:
Patient Report Outcome Measurement | Baseline, 12 weeks, 24 weeks, 36 weeks
  Quality of life based on Physical, Emotional, and Substance Use
Multidimensional Psychological Flexibility Inventory (MPFI) | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  psychological flexibility of behavior, feelings and emotions
CHRONIC PAIN ACCEPTANCE QUESTIONNAIRE | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Feelings of pain and whether they can be accepted or tolerated
AAQ-SA | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Substance use urges and psychological flexibility when it comes to misuse
Mood Symptoms | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Mood symptoms will be assessed by the Patient Health Questionnaire Beck Depression Inventory
Anxiety Symptoms | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Anxiety symptoms will be assessed by the Beck Anxiety Index
Pain catastrophizing | Baseline, 12 weeks, 36 weeks
  Pain catastrophizing will be assessed via the Pain Catastrophizing Scale.
Trauma | Baseline and 24 weeks
  Trauma will be assessed for via the Life Events Checklist.
Opioid craving | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Opioid craving will be assessed for via the Medication Craving Scale.
Substance Use | Baseline, 30 days, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Substance use other than opioid use will be assessed via the ASI
Alcohol Use | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Audit C
Substance use | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  urine toxicology tests.
Anhedonia | Baseline, 24 weeks, 36 weeks
  Anhedonia will be assessed via the Snaith-Hamilton Pleasure Scale (SHAPS).
Sleep | Baseline, 12 weeks, 24 weeks, 36 weeks
  Sleep will be assessed via PROMIS Sleep Disturbance 6a + Sleep Duration Question.
Perceived Stress | Baseline, 12 weeks, 24 weeks, 36 weeks
  NIH Toolbox Perceived Stress Fixed Form 18+.
Stress | Baseline and 24 weeks
  Stress will be assessed via the Urban Life Stress Scale.
Stigma & discrimination | Baseline
  Stigma and discrimination will be assessed via the Perceived discrimination: Everyday discrimination scale.
Suicidality | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Suicidality will be assessed via the Columbia Suicide Severity Rating Scale. CSSR-S
Satisfaction with Therapy | 12 weeks
  Satisfaction with therapy will be assessed by administration of a 13-item 'Satisfaction With Therapy Scale Revised' questionnaire. Responses to the items on the questionnaire will assess the participants' agreement to the various statements that best describe the ACT therapy received over the past 12 weeks based on a 5 point scale ranging from 1 ("Strongly disagree") to 5 ("Strongly agree") for an overall possible score of 13-65 with higher scores denoting increased satisfaction. Group scores will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Perez, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center; Tiffany Liu, MD, Study Director — Montefiore; Brianna Norton, DO, Study Director — Montefiore
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No